CLINICAL TRIAL: NCT07235982
Title: Comparative Study Between Shoulder Anterior Capsular Block Plus Steroid Injection Versus Steroid Injection Alone for Pain Management in Adhesive Capsulitis: A Randomized Trial
Brief Title: Shoulder Anterior Capsular Block and Intraarticular Steroid Injection Versus Intraarticular Steroid Injection for Enhancing Pain Relief in Adhesive Capsulitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Dina Abdelhameed Elsadek Salem, principle investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1593
Record Dates: First submitted 2025-09-29; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Analgesia
Keywords: shoulder anterior capsular block; intraarticular steroid injection; adhesive capsulitis
MeSH Terms: conditions — Agnosia; Bursitis

STUDY DESIGN:
Intervention Model Description: pain relief in adhesive capsulitis by comparing shoulder anterior capsular block and intraarticular steroid injection versus intraarticular steroid injection
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors are blind to the study groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Shoulder anterior capsular block (SHAC) (Active Comparator): patients will receive ultrasound guided (SHAC) block combined with intraarticular steroid injection of the affected shoulder joint
  Interventions: Procedure: Group Group Shoulder anterior capsular block (SHAC)
- Group intraarticular steroid injection (IASI) (Active Comparator): patients will receive intraarticular steroid injection of the affected shoulder joint
  Interventions: Procedure: Group intraarticular steroid injection (IASI)

INTERVENTIONS:
Procedure: Group Group Shoulder anterior capsular block (SHAC) — patients will receive ultrasound guided (SHAC) block combined with intraarticular steroid injection of the affected shoulder joint followed by home exercise program.
  Arms: Group Shoulder anterior capsular block (SHAC)
Procedure: Group intraarticular steroid injection (IASI) — patients will receive intraarticular steroid injection of the affected shoulder joint followed by home exercise program
  Arms: Group intraarticular steroid injection (IASI)

SUMMARY:
Improving pain in the patients with adhesive capsulitis by comparing the effect of combined shoulder anterior capsular block and intraarticular steroid injection versus intraarticular steroid injection.

DETAILED DESCRIPTION:
Comparing between combined shoulder anterior capsular block and intraarticular steroid injection versus intraarticular steroid injection for enhancing pain relief in adhesive capsulitis as regards:

* To measure analgesic parameters including: assessment of pain score by using Visual Analogue Score during 8 weeks follow up in comparison to baseline and total amount of rescue analgesic (ibuprofen) consumption.
* To assess the Shoulder pain and Disability Index
* To record complications of the block (local anesthetic toxicity, infection, bleeding, nerve injury)
* Over all patient's satisfaction: The patients will be asked to rate the overall degree of satisfaction of the analgesia by using a 5-points likert-like verbal scale (1 = very dissatisfied analgesia, 2 = dissatisfied analgesia, and 3 = neutral, 4=satisfied analgesia, and 5=very satisfied analgesia).

ELIGIBILITY:
Inclusion Criteria:

* Patients acceptance
* Age: 41-65 years old
* Sex: both sex (males or females).
* Physical status: American Society of Anesthesiologist (ASA) І, II.
* Patients attend orthopedic or pain clinic with complaint of shoulder pain and stiffness. These patients received conservative management of pain with no relief of symptoms for at least 2 weeks.

Exclusion Criteria:

* Shoulder pain due to secondary causes, e.g. acute trauma, fractures, bony deformity, glenohumeral joint pathology, acromioclavicular joint pathology and rotator cuff disorder.

  * Patient with any contraindications of regional blocks (as coagulopathy or local infection at injection site)
  * Patients with known history of allergy to the study drugs (bupivacaine and methylprednisolone).
  * Advanced hepatic, renal, cardiovascular, neurologic and respiratory diseases, uncontrolled diabetes mellitus and thyroid.
  * History of neuropathy in the involved limb or previous revision surgery.

Ages: 41 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
pain intensity | BEFORE STARTING PROCEDURE (0 hour)(baseline)
  measured by Visual Analogue Scale (VAS) 10 cm line labelled (0-10), in which 0 presents no pain and 10 represents the worst pain in each participant
pain intensity | 15 minutes after the procedure
  measured by Visual Analogue Scale(VAS) as 10 cm line labelled (0-10), in which 0 presents no pain and 10 represents the worst pain in each participant
pain intensity | first 6 hours postoperative
  measured by Visual Analogue Scale (VAS) 10 cm line labelled (0-10), in which 0 presents no pain and 10 represents the worst pain in each participant
pain intensity | one week after procedure
  measured by Visual Analogue Scale (VAS) 10 cm line labelled (0-10), in which 0 presents no pain and 10 represents the worst pain in each participant
pain intensity | 3 weeks after procedure
  measured by Visual Analogue Scale (VAS) 10 cm line labelled (0-10), in which 0 presents no pain and 10 represents the worst pain in each participant
pain intensity | 6 weeks after procedure
  measured by Visual Analogue Scale (VAS) 10 cm line labelled (0-10), in which 0 presents no pain and 10 represents the worst pain in each participant
pain intensity | 8 weeks after procedure
  measured by Visual Analogue Scale (VAS) 10 cm line labelled (0-10), in which 0 presents no pain and 10 represents the worst pain in each participant

SECONDARY OUTCOMES:
Assessment of Shoulder Pain and Disability Index (SPADI) | baseline (0 ) and subsequently at one week, 3 weeks , 6 weeks and 8 weeks after procedure
  SPADI contains 13 items that assess two domains - a five item subscale that measures pain and an eight item subscale that measures disability. Each subscale scored 10 ranging from 0 (best) to 10 (worst). It is a self administered, valid questionnaire,
Total amount of rescue analgesia | first 24 hours
  Total amount of rescue analgesia (ibuprofen)
patient's satisfaction | 1 week after procedure
  degree of satisfaction of the analgesia by using a 5-points likert-like verbal scale (1 = very dissatisfied analgesia, 2 = dissatisfied analgesia, and 3 = neutral, 4=satisfied analgesia, and 5=very satisfied analgesia)
Complications of SHAC block | 24 hours
  Complications of SHAC block (local anesthetic toxicity, infection, bleeding)
PASSIVE AND ACTIVE RANGE OF MOTION | at baseline, first week and third week follow up post intervention.
  Passive and active shoulder flexion, abduction, and external rotation will be measured using goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Dina Salem, MD, Principal Investigator — FACULTY OF MEDICINE, ZAGAZIG UNIVERSITY
Locations (1):
- Faculity of Medicine, Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No